CLINICAL TRIAL: NCT03424603
Title: A Phase 1 Open-Label, Safety, Pharmacokinetic and Preliminary Efficacy Study of STRO-001, an Anti-CD74 Antibody Drug Conjugate, in Patients With Advanced B-Cell Malignancies
Brief Title: Study of STRO-001, an Anti-CD74 Antibody Drug Conjugate, in Patients With Advanced B-Cell Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sutro Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STRO-001-BCM1
Record Dates: First submitted 2018-01-24; First posted 2018-02-07 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: B-cell Lymphoma; Non Hodgkin Lymphoma; Multiple Myeloma; Follicular Lymphoma; Mantle Cell Lymphoma; Diffuse Large B Cell Lymphoma; Indolent Lymphoma; B Cells--Tumors
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Multiple Myeloma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- STRO-001 (Experimental): intravenous
  Interventions: Drug: STRO-001

INTERVENTIONS:
Drug: STRO-001 — intravenous antibody drug conjugate

SUMMARY:
First-in-human Phase 1 trial to study the safety, pharmacokinetics and preliminary efficacy of STRO-001 given intravenously every 3 weeks.

DETAILED DESCRIPTION:
This study is a first-in-human Phase 1, open-label, multicenter, dose escalation study with dose expansion to identify the maximum tolerated dose (MTD), the recommended phase 2 doses (RP2D) and to evaluate the safety, tolerability, and preliminary anti-tumor activity of STRO-001 in adult subjects with B-cell malignancies (MM and NHL) who are refractory to, or intolerant of, all established therapy known to provide clinical benefit for their condition (i.e., trial subjects must not be candidates for any regimens known to provide clinical benefit). The study will consist of two parts: Part 1, dose escalation, and Part 2, dose expansion.

The study uses an accelerated dose titration design for dose escalation. Doses will be escalated using an N-of-1 per dosing cohort until the first instance of a treatment-related, clinically relevant Grade 2 non-hematologic toxicity or a Grade 3 hematologic toxicity of any type is observed during Cycle 1 (first 21 days). Following this a standard 3+3 trial design is used for all further escalation cohorts. Dose escalation is conducted independently for the two dose escalation tumor cohorts (MM and NHL). A recommended STRO-001 dose for expansion will be determined for MM and NHL.

The dose expansion (Part 2) portion of the study will begin when Part 1 is completed. Enrollment in dose expansion will include separate tumor cohorts of MM and NHL.

In both Part 1 and Part 2 of the study, STRO-001 will be dosed as an intravenous (IV) infusion on Day 1 of a 21-day cycle, until disease progression. Labs will be drawn on a weekly basis for Cycles 1-4, and every three weeks starting with Cycle 5. Weekly clinical evaluations will be conducted during the first 4 cycles; thereafter, clinical evaluations will be conducted on infusion days (Day 1 of each cycle). Samples for pharmacokinetics (PK) analysis will occur at specific times on Days 1, 2, and 8 of the first two cycles of treatment, Day 1 of the third cycle of treatment and at End of Treatment visit. Additional clinical evaluations and labs may occur at the discretion of the investigator.

Subjects who receive any dose of STRO-001 will be included in safety analyses. Disease evaluations will include peripheral blood analysis, bone marrow assessments and scans as appropriate. Disease status will be evaluated per MM-specific or NHL-specific criteria. Samples will be collected to assess the PK and immunogenicity of STRO-001. Biomarkers may be assessed from bone marrow, peripheral blood and/or tissue samples. Subjects will continue to receive study drug until disease progression, unacceptable toxicity, withdrawal of consent, or end of study (study completion).

ELIGIBILITY:
Key Inclusion Criteria:

1. Confirmation of diagnosis
2. Relapsed or relapsed/refractory disease
3. Age ≥ 18 years
4. ECOG performance status (0-2)
5. Life expectancy > 3 months
6. Adequate bone marrow and renal functions
7. QTcF <500 msec
8. Ability to comply with treatment, PK and test schedules
9. NHL only- at least one measurable lesion

Key Exclusion Criteria:

1. Active plasma cell leukemia and/or leukemic manifestations of lymphoma
2. Known amyloidosis (MM patients)
3. Chronic lymphocytic leukemia and Richter's transformation, and prolymphocytic leukemia (NHL subjects)
4. T-cell malignancy
5. Sensory or motor neuropathy ≥ grade 2
6. Chronic or ongoing active infectious disease requiring systemic treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis and active hepatitis C
7. Ongoing immunosuppressive therapy, including systemic corticosteroids. Note: Subjects may be using topical or inhaled corticosteroids.
8. Clinically significant cardiac disease
9. Significant concurrent, uncontrolled medical condition
10. History or clinical signs of meningeal or active CNS involvement
11. Known severe chronic obstructive pulmonary disease or asthma
12. History of significant cerebrovascular disease
13. Known Human Immunodeficiency Virus seropositivity
14. Positive serology for hepatitis B defined by a positive test for HBsAg
15. Concurrent participation in another therapeutic treatment trial
16. High screening liver function tests
17. Prior treatment with CD74 targeting therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Part 1: Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability of STRO-001) | 18 months
  Incidence of adverse events (AEs) observed across STRO-001 dose levels
Part 1: Define the recommended phase 2 dose (RP2D) and maximum tolerated dose (MTD) of STRO-001 | 18 months
  Frequency of dose-limiting toxicity and exposure across STRO-001 dose levels
Part 2: Evaluate preliminary anti-tumor activity (multiple myeloma patients) | 24 months
  Objective response rates per International Myeloma Working Group (IMWG) criteria for response assessment
Part 2: Evaluate preliminary anti-tumor activity (NHL patients) | 24 months
  Objective response rates per the Lugano classification for response assessment

SECONDARY OUTCOMES:
Part 1: Characterize the pharmacokinetics (PK) of STRO-001 by measuring the maximum plasma concentration (Cmax) | 18 months
  Measurement of maximum plasma concentration after the administration of STRO-001
Part 1: Characterize the PK of STRO-001 by measuring the half-life (t1/2) of STRO-001 | 18 months
  Measurement of terminal half-life of STRO-001 after the administration of STRO-001
Part 1: Characterize the PK of STRO-001 measuring the total area under the concentration versus time curve from zero to infinity (AUCinf) | 18 months
  Measurement of AUC to infinity (AUCinf)
Part 1: Characterize the PK of STRO-001 by measuring the clearance (CL) | 18 months
  Measurement of total body clearance
Part 1: Characterize the PK of STRO-001 by measuring the the steady state volume of distribution (Vss) | 18 months
  Measurement of steady state volume of distribution
Part 1: Assess the immunogenic potential of STRO-001 | 18 months
  Evaluation and quantitation of circulating anti-drug antibodies (ADAs) over time
Part 2: Further evaluate the incidence of Treatment-Emergent Adverse Events (Safety and Tolerability of STRO-001) | 24 months
  Number of patients with abnormal laboratory values and/or adverse events related to STRO-001 treatment
Part 2: Evaluate preliminary anti-tumor efficacy with a time-to-event analysis of duration of response (DOR) in patients treated with STRO-001 | 24 months
  Each cohort will be analyzed independently
Part 2: Evaluate preliminary anti-tumor efficacy with a time-to-event analysis of progression-free survival (PFS) in patients treated with STRO-001 | 24 months
  Each cohort will be analyzed independently
Part 2: Characterize the PK of STRO-001 by measuring the maximum plasma concentration (Cmax) | 24 months
  Measurement of maximum plasma concentration after the administration of STRO-001
Part 2: Characterize the PK of STRO-001 by measuring the half-life (t1/2) of STRO-001 | 24 months
  Measurement of terminal half-life of STRO-001 after the administration of STRO-001
Part 2: Characterize the PK of STRO-001 by measuring the area under the plasma concentration versus time curve (AUC) | 24 months
  Measurement of AUC to infinity (AUC inf)
Part 2: Characterize the PK of STRO-001 by measuring the clearance (CL) | 24 months
  Measurement of total body clearance

OTHER OUTCOMES:
Part 1: Preliminary assessment of the anti-tumor activity of STRO-001 (multiple myeloma patients) | 18 months
  Objective response rates per IMWG criteria for response assessment
Part 1: Preliminary assessment of the anti-tumor activity of STRO-001 (NHL) | 18 months
  Objective response rates per the Lugano classification for response assessment (NHL patients)

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Molina, MD, Study Director — Sutro Biopharma
Locations (22):
- United States (22):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Oncology Associates, PC--HOPE Division, Tucson, Arizona
  - City of Hope Medical Center, Duarte, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Univeristy of California San Francisco HDF Comprehensive Cancer Center, San Francisco, California
  - Rocky Mountain Cancer Center, Aurora, Colorado
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Kansas Cancer Center, Fairway, Kansas
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Cancer Institute, Detroit, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Texas Oncology, Austin, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - UT Health San Antonio, San Antonio, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - West Virginia University, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: ASH conference, Dec 2017 oral presentation NHL abstract — https://ash.confex.com/ash/2017/webprogram/Paper102382.html
- See also: ASH conference, Dec 2017 poster presentation multiple myeloma abstract — https://ash.confex.com/ash/2017/webprogram/Paper104213.html